CLINICAL TRIAL: NCT02665286
Title: Methocarbamol and Orphenadrine for Acute, Non-traumatic, Non-radicular Low Back Pain: A Randomized, Placebo Controlled, 3-armed Study
Brief Title: Orphenadrine and Methocarbamol for LBP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Associate Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-5903
Record Dates: First submitted 2016-01-15; First posted 2016-01-27 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Orphenadrine; Cholinergic Antagonists; Methocarbamol; Naproxen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Naproxen 500mg tablets taken twice per day + placebo. Placebo dose will be either 1 capsule orally twice per day or 1 or 2 capsules orally, thrice per day Naproxen 500mg po BID x 10 days #20 + Placebo
  Interventions: Drug: Naproxen; Drug: Placebo
- Orphenadrine (Active Comparator): Naproxen 500mg, orally twice per day + orphenadrine 100mg, orally twice per day for 10 days Naproxen 500mg po BID x 10 days #20 + Orphenadrine
  Interventions: Drug: Orphenadrine; Drug: Naproxen
- Methocarbamol (Active Comparator): Naproxen 500mg tablets, orally twice per day + methocarbamol 750mg, orally as 1 or 2 tabs, thrice per day Naproxen 500mg po BID x 10 days #20 + Methocarbamol
  Interventions: Drug: Methocarbamol; Drug: Naproxen

INTERVENTIONS:
Drug: Orphenadrine — Orphenadrine 100mg PO BID x 7 days
  Other Names: anticholinergic drug
  Arms: Orphenadrine
Drug: Methocarbamol — Methocarbamol 750mg 1-2 tabs po TID x 7 days
  Other Names: Muscle relaxant
  Arms: Methocarbamol
Drug: Naproxen — Naproxen 500mg PO BID x 7 days
  Other Names: nonsteroidal anti-inflammatory drug
Drug: Placebo — 1/2 of placebo packages will be dosed to match methocarbamol: 1-2 tabs po TID x 7days 1/2 of placebo packages will be dosed to match orphenadrine: 1 tab PO BID x 7 days
  Arms: Placebo

SUMMARY:
Low back pain is a common cause of visit to emergency department. It is not clear if skeletal muscle relaxants are of benefit for patients with acute low back pain. This is a randomized study to determine if skeletal muscle relaxants, when combined with naproxen, improve outcomes more than naproxen alone

DETAILED DESCRIPTION:
Patients with acute, non-traumatic, non-radicular low back pain will be enrolled at the time of discharge from the emergency department. Participants will be followed by telephone one week and 3 months after the ED visit

ELIGIBILITY:
Inclusion Criteria:

* LBP duration <= 2 weeks
* No trauma to low back within previous month
* No radicular symptoms
* No history of low back pain or history of only infrequent episodes

Exclusion Criteria:

* Medication allergies or contra-indications
* Not available for follow-up
* Chronic pain syndrome

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Friedman, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Friedman BW, Cisewski D, Irizarry E, Davitt M, Solorzano C, Nassery A, Pearlman S, White D, Gallagher EJ. A Randomized, Double-Blind, Placebo-Controlled Trial of Naproxen With or Without Orphenadrine or Methocarbamol for Acute Low Back Pain. Ann Emerg Med. 2018 Mar;71(3):348-356.e5. doi: 10.1016/j.annemergmed.2017.09.031. Epub 2017 Oct 28. PMID 29089169

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Naproxen 500mg po BID x 10 days #20 + Placebo
  Naproxen: Naproxen 500mg PO BID x 7 days
  Placebo: 1/2 of placebo packages will be dosed to match methocarbamol: 1-2 tabs po TID x 7days 1/2 of placebo packages will be dosed to match orphenadrine: 1 tab PO BID x 7 days
- Orphenadrine: Naproxen 500mg po BID x 10 days #20 + Orphenadrine
  Orphenadrine: Orphenadrine 100mg PO BID x 7 days
  Naproxen: Naproxen 500mg PO BID x 7 days
- Methocarbamol: Naproxen 500mg po BID x 10 days #20 + Methocarbamol
  Methocarbamol: Methocarbamol 750mg 1-2 tabs po TID x 7 days
  Naproxen: Naproxen 500mg PO BID x 7 days
Period: Overall Study
Arm/Group | Placebo | Orphenadrine | Methocarbamol
Started | 79 | 80 | 81
Completed | 76 | 78 | 80
Not Completed | 3 | 2 | 1
Not completed — Lost to Follow-up | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Orphenadrine | Methocarbamol | Total
Number analyzed (Participants) | 79 | 80 | 81 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (12) | 40 (12) | 38 (12) | 39 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 41 | 109
  Male | 45 | 46 | 40 | 131
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 79 | 80 | 81 | 240
Duration of Back Pain Prior to Study [Median (Inter-Quartile Range); unit: Hours] | 48 [24 to 108] | 72 [24 to 96] | 48 [24 to 120] | 48 [24 to 96]

OUTCOME MEASURES:

1. Primary Outcome: Functional Impairment as Measured on the Roland Morris Disability Questionnaire
Description: Change in Roland Morris Disability Questionnaire between baseline and 1 week.
  The low back pain functional disability scale is the RMDQ. The RMDQ is a 24-item low back pain functional scale recommended for use in low back pain research.Higher scores signify greater low back-related functional impairment.0= no functional impairment, 24= severe functional impairment.
Time Frame: 1 week
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Orphenadrine | Methocarbamol
Number analyzed (Participants) | 76 | 78 | 80
units on a scale | 10.9 [8.9 to 12.9] | 9.4 [7.4 to 11.5] | 8.1 [6.1 to 10.1]

2. Secondary Outcome: Cases of Moderate or Severe LBP
Description: Participants with moderate to severe low back pain after treatment as report on the following ordinal scale: severe, moderate, mild, or none
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Orphenadrine | Methocarbamol
Number analyzed (Participants) | 76 | 78 | 80
Participants | 34 | 26 | 31

3. Secondary Outcome: Medications--Patient Self Report of Medication Use
Description: Participants still using medication such as analgesics for LBP after treatment
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Orphenadrine | Methocarbamol
Number analyzed (Participants) | 76 | 78 | 80
Participants | 42 | 40 | 50

4. Secondary Outcome: Patient Satisfaction With Treatment
Description: The number of participants with affirmative response to the following question: Do you want the same medication combination during a subsequent episode of LBP. This is a patient-centered outcome that allows each individual to determine the desirability of the intervention.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Orphenadrine | Methocarbamol
Number analyzed (Participants) | 75 | 78 | 78
Participants | 51 | 53 | 51

ADVERSE EVENTS:
Time Frame: 1 week after treatment
Arm/Group | Placebo | Orphenadrine | Methocarbamol
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/78 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/78 | 0/80
Other Adverse Events (participants affected / at risk) | 9/76 | 8/78 | 14/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Orphenadrine (N=78) | Methocarbamol (N=80)
Drowsy (Nervous system disorders) | 5 (5) | 8 (8) | 13 (13)
dizz (Nervous system disorders) | 2 (2) | 3 (3) | 4 (4)
Stomach irritation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT02665286/Prot_SAP_000.pdf